CLINICAL TRIAL: NCT06668025
Title: Application of Myxovirus Resistance Protein a in Antiviral Treatment Guidance of Respiratory Viral Infections
Brief Title: MxA-Guided Antiviral Treatment in Respiratory Viral Infections
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Capital Medical University (Other)
Collaborators: China-Japan Friendship Hospital (Other); Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bin Cao, Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2023-I2M-C&T-B-119
Record Dates: First submitted 2024-10-30; First posted 2024-10-31 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2024-10

CONDITIONS: Respiratory Viral Infections; Influenza; SARS CoV-2
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MxA group (Experimental): Perform MxA test; MxA results reported to attending clinicians; Provide MxA-based guidelines on antiviral treatment to attending clinicians; Telephone Visit at Day 30
  Interventions: Other: MxA tests; Other: MxA feedback; Other: Follow-up at Day 30
- Control group (Active Comparator): Telephone Visit at Day 30
  Interventions: Other: Follow-up at Day 30

INTERVENTIONS:
Other: MxA tests — Whole blood samples will be collected on Days 1, 4, 7, and 10 for MxA testing. MxA measurements on Days 4, 7, and 10 will be performed only for patients still hospitalized on antiviral thearpy or at the attending physician's discretion.
  Arms: MxA group
Other: MxA feedback — MxA results will be reported to the attending physician within 4 hours, along with MxA-based antiviral treatment guidelines.
  Arms: MxA group
Other: Follow-up at Day 30 — A telephone visit will be conducted on or around Day 30 for study participants who are discharged, to collect information on antiviral usage, recurrence infection, readmissions, and additional medical visits.

SUMMARY:
This pilot randomized controlled trial (RCT) will investigate the clinical impact of Myxovirus Resistance Protein A (MxA)-guided antiviral treatment versus standard treatment in patients with respiratory viral infections.

DETAILED DESCRIPTION:
Effective antiviral treatment would shorten the time to symptom resolution, accelerate the cessation of viral shedding, and improve the prognosis of respiratory viral infections. However, the optimal timing for antiviral treatment remains undetermined, and the current lack of objective biomarkers for respiratory viral infections often leads to either prolonged or insufficient antiviral treatment. Thus, there is a need for strategies that incorporate novel diagnostics to guide antiviral treatment and provide more individualized therapy.

Myxovirus resistance protein A (MxA), a novel marker of viral infection, may hold potential in guiding antiviral therapy. In this pilot randomized controlled clinical study, we aim to evaluate whether MxA-guided antiviral treatment, as compared to standard care, can reduce the recurrence rate of respiratory viral infections and improve clinical outcomes

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years old
* With a primary diagnosis of influenza or COVID-19 infection, diagnosed by a rapid antigen test or RT-PCR
* Duration of infection ≤14 days for non-severe patients and < 28 days for patients with severe infections
* Currently receiving or planned to receive antiviral treatment, with the attending physician yet to decide on the discontinuation of the antiviral treatment

Exclusion Criteria:

* Current endotracheal intubation and mechanical ventilation
* Current vasopressor use
* Known immunosuppression
* Received interferon therapy within 30 days before screening
* Systemic inflammatory responses within 30 days prior to screening, such as cerebral infarction, myocardial infarction, or surgery
* Received vaccine in the past 30 days
* Active tuberculosis
* With contraindications for antiviral treatment
* Unable to obtain eligible samples
* Co-infected with influenza and COVID-19

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
30-Day recurrence rate | 30 days
  Recurrence is defined as the worsening of symptoms and a positive viral PCR test from respiratory samples in patients who discontinued antiviral treatment within 30 days of enrollment.

SECONDARY OUTCOMES:
Antiviral-days by day 30 | 30 days
  Defined as the total number of days of antiviral treatment from randomization to the discontinuation of antiviral therapy by Day 30.
Length of hospital stay | 30 days
  Defined as the total number of hospital days by Day 30.
30-day mortality | 30 days
  Defined as the proportion of patients who died by Day 30.
Incidence of mechanical ventilation | 30 days
  Defined as the proportion of patients receiving mechanical ventilation by day 30.
Incidence of complications | 30 days
  Defined as the incidence of complications such as bronchitis and viral pneumonia occurring within 30 days of enrollment in patients with an initial diagnosis of upper respiratory viral infection.
ICU admission rate | 30 days
  Defined as the incidence of transfer to the ICU within 30 days of enrollment for patients initially admitted to a general ward.
Readmission rate | 30 days
  Defined as the incidence of readmission or additional medical visits within 30 days of enrollment for patients who have been discharged.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Cao, Study Director — China-Japan Friendship Hospital
Locations (1):
- China-Japan Friendship hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
IPD used in the results publication will be shared.
Supporting Information: ICF, CSR